CLINICAL TRIAL: NCT02386098
Title: A Phase 2b Randomized, Active-Controlled, Staged, Open-Label Trial to Investigate Safety and Efficacy of BMS-955176/GSK3532795 in Combination With Dolutegravir and Atazanavir (With or Without Ritonavir) in Treatment-Experienced HIV-1 Infected Adults
Brief Title: Strategy-confirming Study of BMS-955176 to Treat HIV-1 Infected Treatment-experienced Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: GI Intolerability
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205892; AI468-048 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2015-03-06; First posted 2015-03-11 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — BMS-955176; Atazanavir Sulfate; Ritonavir; dolutegravir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1: BMS-955176 + ATV + RTV + DTG (Experimental): BMS-955176 at 120 mg tablet per day + Atazanavir boosted with ritonavir (ATV/r) 300/100 mg tablets per day + DTG 50 mg tablet per day, orally
  Interventions: Drug: BMS-955176; Drug: Atazanavir (ATV); Drug: Ritonavir (RTV); Drug: Dolutegravir (DTG)
- Arm 2: TDF + ATV + RTV + DTG (Other): TDF 300 mg tablet per day + ATV/r at 300/100 mg tablets per day + DTG 50 mg per day, orally
  Interventions: Drug: Atazanavir (ATV); Drug: Ritonavir (RTV); Drug: Dolutegravir (DTG); Drug: Tenofovir (TDF)
- Arm 3: BMS-955176 + ATV + DTG (Experimental): BMS-955176 at 120 mg tablet per day + ATV at 400 mg tablet per day + DTG at 50 mg tablet per day, orally
  Interventions: Drug: BMS-955176; Drug: Atazanavir (ATV); Drug: Dolutegravir (DTG)
- Arm 4: BMS-955176 + ATV + DTG (Experimental): BMS-955176 at 180 mg tablet per day + ATV at 400 mg tablet per day + DTG at 50 mg tablet per day, orally
  Interventions: Drug: BMS-955176; Drug: Atazanavir (ATV); Drug: Dolutegravir (DTG)
- Arm 5: TDF + ATV + RTV + DTG (Other): TDF 300 mg tablet per day + ATV/r at 300/100 mg tablets per day + DTG 50 mg per day, orally
  Interventions: Drug: Atazanavir (ATV); Drug: Ritonavir (RTV); Drug: Dolutegravir (DTG); Drug: Tenofovir (TDF)

INTERVENTIONS:
Drug: BMS-955176 — HIV Maturation Inhibitor
  Arms: Arm 1: BMS-955176 + ATV + RTV + DTG; Arm 3: BMS-955176 + ATV + DTG; Arm 4: BMS-955176 + ATV + DTG
Drug: Atazanavir (ATV) — Atazanavir
Drug: Ritonavir (RTV) — Ritonavir
  Arms: Arm 1: BMS-955176 + ATV + RTV + DTG; Arm 2: TDF + ATV + RTV + DTG; Arm 5: TDF + ATV + RTV + DTG
Drug: Dolutegravir (DTG) — Dolutegravir
Drug: Tenofovir (TDF) — Tenofovir
  Arms: Arm 2: TDF + ATV + RTV + DTG; Arm 5: TDF + ATV + RTV + DTG

SUMMARY:
The purpose of this study is to evaluate whether the combination of BMS-955176 with atazanavir (ATV) [with or without ritonavir (RTV)] and dolutegravir (DTG) is efficacious, safe, and well-tolerated in HIV-1 infected treatment experienced adults.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women, at least 18 years of age
* Antiretroviral treatment-experienced, defined as having documented evidence of having failed 1 or 2 regimens that include 2 or 3 classes of antiretroviral (ARV) (with or without documented resistance)
* CD4+ T-cell count > 50 cells/mm3
* Screening genotype/phenotype indicating susceptibility to study drugs (unboosted ATV, FC < 2.2; DTG; TDF)

Exclusion Criteria:

* Antiretroviral treatment-experienced adults who have failed > 2 ARV regimens
* Resistance or partial resistance to any study drug determined by tests at Screening
* Historical or documented genotypic and/or phenotypic drug resistance testing showing certain resistance mutations to ATV, TDF, RAL, Protease Inhibitors, and certain TAMs
* Chronic hepatitis B virus (HBV)/ hepatitis C virus (HCV)
* Blood tests that indicate normal liver function
* Hemoglobin < 8.0 g/dL, Platelets < 50,000 cells/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (54):
- United States (16):
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
- Argentina (5):
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Mar del Plata
- Australia (3):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Darlinghurst, Sydney, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
- Canada (4):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Chile (3):
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Providencia, Santiago de Chile
  - GSK Investigational Site, Santiago
- Colombia (3):
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Cali
- Mexico (6):
  - GSK Investigational Site, Juárez, Chihuahua
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, DF
  - GSK Investigational Site, Distrito Federal
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Oaxaca City
- GSK Investigational Site, Lima, Peru
- GSK Investigational Site, San Juan, Puerto Rico
- Russia (5):
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Yekaterinburg
- South Africa (4):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Bloemfontein, Free State
  - GSK Investigational Site, Tembisa
  - GSK Investigational Site, Westdene
- Taiwan (2):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taipei
- GSK Investigational Site, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was planned to be conducted in two Stages (96 weeks each); but was terminated early during Stage 1 due to high rates of gastrointestinal (GI) intolerability and early end of the concurrent, 205891 (NCT02415595) formal dose-finding study. Hence, data was collected only in Stage 1 and no participants were enrolled in Stage 2.
Pre-assignment Details: A total of 288 participants were screened, of which 86 were randomized in a ratio of 1:1 to one of the two treatment arms in Stage 1.
Groups:
- Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD: Participants were administered a once daily (QD) oral dose of 120 milligram (mg) BMS-955176 in combination with atazanavir boosted with ritonavir (ATV/r) 300/100 mg QD and dolutegravir (DTG) 50 mg QD for a duration of 96 weeks. The doses were administered in the morning with a meal.
- Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD: Participants were administered a QD oral dose of 300 mg tenofovir (TDF) in combination with ATV/r 300/100 mg QD and DTG 50 mg QD for a duration of 96 weeks. The doses were administered in the morning with a meal.
- Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD: Participants were planned to be administered a QD oral dose of 120 mg BMS-955176 in combination with atazanavir without ritonavir (ATV) 400 mg QD and DTG 50 mg QD for a duration of 96 weeks.
- Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD: Participants were planned to be administered a QD oral dose of 180 mg BMS-955176 in combination with ATV 400 mg QD and DTG 50 mg QD for a duration of 96 weeks.
- Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD: Participants were planned to be administered a QD oral dose of 300 mg TDF in combination with ATV/r 300/100 mg QD and DTG 50 mg QD for a duration of 96 weeks.
Period: Stage 1 (96 Weeks)
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Started | 43 | 43 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 43 | 43 | 0 | 0 | 0
Not completed — Other: Administrative reason by sponsor | 30 | 29 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0 | 0 | 0
Not completed — Other:Protocol defined stopping criteria | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0
Not completed — Other: Breach of good clinical practice | 5 | 8 | 0 | 0 | 0
Period: Stage 2 (96 Weeks)
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Started | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent to treat (mITT) Population comprised of randomized participants who received at least one dose of BMS-955176 or TDF. Data from 13 participants randomized at a single site were excluded due to a breach of good clinical practice (GCP) that indicated participants may not have been properly consented to participate in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Total
Number analyzed (Participants) | 38 | 35 | 0 | 0 | 0 | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.8 (11.45) | 41.7 (12.06) |  |  |  | 40.7 (11.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 |  |  |  | 15
  Male | 31 | 27 |  |  |  | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 17 |  |  |  | 31
  Black/African American | 6 | 2 |  |  |  | 8
  Asian | 4 | 4 |  |  |  | 8
  Unknown | 14 | 12 |  |  |  | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) <40 Copies Per Milliliter (c/mL) at Week 24-Stage 1
Description: Blood samples were collected for quantitative analysis of plasma HIV-1 RNA. Percentage of participants with plasma HIV-1 RNA <40 c/mL at Week 24 was assessed using the Food and Drug Administration (FDA) snapshot algorithm which used the last on-treatment plasma HIV-1 RNA measurement, within an FDA-specified visit window (18 to 30 weeks), to determine response. Analysis was performed on the modified intent to treat (mITT) Population which comprised of all randomized participants who received atleast one dose of BMS-955176 or TDF.
Time Frame: Week 24
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 38 | 35
Percentage of participants | 73.7 [56.9 to 86.6] | 60.0 [42.1 to 76.1]

2. Primary Outcome: Percentage of Participants With Plasma HIV-1 RNA <40 c/mL at Week 24-Stage 2
Description: Blood samples were planned to be collected for quantitative analysis of plasma HIV-1 RNA. The analysis was not performed in Stage 2 due to early termination of the study during Stage 1.
Time Frame: Week 24
Population: mITT Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <40 c/mL at Weeks 48 and 96-Stage 1
Description: Blood samples were collected for quantitative analysis of plasma HIV-1 RNA. Response was assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a participant's response status. The percentage of responders with HIV-1 RNA <40 c/mL at Weeks 48 and 96 using mITT Population (observed) which consisted of participants in the mITT Population excluding participants who had no HIV-1 RNA result data in the assessment visit windows due to discontinuation and who discontinued on or after the date of site notification of study termination by the sponsor (October 10, 2016) is presented. The study was terminated early during the primary end point analysis of Stage 1; hence, data was not collected for Week 96 analysis.
Time Frame: Weeks 48 and 96
Population: mITT Population (observed). Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 38 | 35
Percentage of participants
  Week 48; n=8, 9: number analyzed (Participants) | 8 | 9
  Week 48; n=8, 9 | 75.0 [34.9 to 96.8] | 66.7 [29.9 to 92.5]
  Week 96; n=0, 0: number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <40 c/mL at Weeks 48 and 96-Stage 2
Description: as for outcome 2
Time Frame: Weeks 48 and 96
Population: mITT Population (observed). Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA <200 c/mL at Weeks 24, 48 and 96-Stage 1
Description: Blood samples were collected for quantitative analysis of plasma HIV-1 RNA. Response was assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a participant's response status. The percentage of responders with HIV-1 RNA <200 c/mL at Weeks 24, 48 and 96 using mITT Population (observed) which consisted of participants in the mITT Population excluding participants who had no HIV-1 RNA result data in the assessment visit windows due to discontinuation and who discontinued on or after the date of site notification of study termination by the sponsor (October 10, 2016) is presented. The study was terminated early during the primary end point analysis of Stage 1; hence, data was not collected for Week 96 analysis.
Time Frame: Weeks 24, 48 and 96
Population: mITT Population (observed). Only those participants with data available at specified time points were analyzed (indicated by n=X in category titles)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 38 | 35
Percentage of participants
  Week 24; n=32, 29: number analyzed (Participants) | 32 | 29
  Week 24; n=32, 29 | 93.8 [79.2 to 99.2] | 89.7 [72.6 to 97.8]
  Week 48; n=8, 9: number analyzed (Participants) | 8 | 9
  Week 48; n=8, 9 | 100 [63.1 to 100.0] | 100 [66.4 to 100.0]
  Week 96; n=0, 0: number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA <200 c/mL at Weeks 24, 48 and 96-Stage 2
Description: as for outcome 2
Time Frame: Weeks 24, 48 and 96
Population: mITT Population (observed). Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Logarithm to the Base 10 (log10) HIV-1 RNA Over Time-Stage 1
Description: Blood samples were collected for analysis of HIV-1 RNA. Baseline is the last value on or before the start of study treatment. Change from Baseline was calculated as the value at specified visit minus the Baseline value. Change from Baseline in plasma HIV-1 RNA (log10) is summarized over time for the mITT Population using observed values, which excluded participants without HIV-1 RNA result data in the assessment visit windows due to discontinuation and who discontinued on or after the date of site notification of study termination by the sponsor (10 October 2016). NA indicates data was not available. The standard deviation could not be calculated as a single participant was analyzed at the specified time point.
Time Frame: Baseline and up to Week 72
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: log10 c/mL
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 38 | 35
log10 c/mL
  Week 2; n=10, 5: number analyzed (Participants) | 10 | 5
  Week 2; n=10, 5 | -4.232 (0.8779) | -4.050 (1.3413)
  Week 4; n=37, 33: number analyzed (Participants) | 37 | 33
  Week 4; n=37, 33 | -4.400 (0.8983) | -3.922 (1.5241)
  Week 8; n=37, 30: number analyzed (Participants) | 37 | 30
  Week 8; n=37, 30 | -4.103 (1.8696) | -4.145 (1.1350)
  Week 12; n=36, 32: number analyzed (Participants) | 36 | 32
  Week 12; n=36, 32 | -4.394 (0.9011) | -4.113 (1.1280)
  Week 16; n=34, 32: number analyzed (Participants) | 34 | 32
  Week 16; n=34, 32 | -4.402 (0.9267) | -4.074 (1.1437)
  Week 24; n=32, 29: number analyzed (Participants) | 32 | 29
  Week 24; n=32, 29 | -4.220 (1.5130) | -4.079 (1.1754)
  Week 32; n=23, 23: number analyzed (Participants) | 23 | 23
  Week 32; n=23, 23 | -4.381 (1.0267) | -3.364 (2.7492)
  Week 40; n=21, 15: number analyzed (Participants) | 21 | 15
  Week 40; n=21, 15 | -4.366 (1.0553) | -4.400 (1.0572)
  Week 48; n=8, 9: number analyzed (Participants) | 8 | 9
  Week 48; n=8, 9 | -4.508 (1.1333) | -4.680 (1.0607)
  Week 60; n=4, 3: number analyzed (Participants) | 4 | 3
  Week 60; n=4, 3 | -5.037 (1.2665) | -4.977 (1.4043)
  Week 72; n=1, 1: number analyzed (Participants) | 1 | 1
  Week 72; n=1, 1 | -3.326 (NA) — The standard deviation could not be calculated as a single participant was analyzed at the specified time point. | -5.713 (NA) — The standard deviation could not be calculated as a single participant was analyzed at the specified time point.

8. Secondary Outcome: Change From Baseline in log10 HIV-1 RNA Over Time-Stage 2
Description: This end point was not evaluated in Stage 2 due to early termination of the study during Stage 1.
Time Frame: Baseline and up to Week 96
Population: mITT Population (observed). Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4+ (CD4+) Cell Count Over Time-Stage 1
Description: The CD4+ cell count was assessed using flow cytometry. Baseline is the last value on or before the start of study treatment. Change from Baseline was calculated as the value at specified visit minus the Baseline value. NA indicates data was not available. The standard deviation could not be calculated as a single participant was analyzed at the specified time point.
Time Frame: Baseline and up to Week 72
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 38 | 35
Cells per microliter
  Week 4; n=37, 33: number analyzed (Participants) | 37 | 33
  Week 4; n=37, 33 | 57.6 (93.54) | 26.7 (83.30)
  Week 8; n=36, 30: number analyzed (Participants) | 36 | 30
  Week 8; n=36, 30 | 77.6 (130.59) | 53.7 (76.57)
  Week 12; n=35, 32: number analyzed (Participants) | 35 | 32
  Week 12; n=35, 32 | 90.4 (190.31) | 115.1 (159.22)
  Week 16; n=34, 31: number analyzed (Participants) | 34 | 31
  Week 16; n=34, 31 | 83.2 (116.78) | 93.8 (113.61)
  Week 24; n=31, 28: number analyzed (Participants) | 31 | 28
  Week 24; n=31, 28 | 127.2 (146.37) | 109.5 (124.35)
  Week 32; n=23, 22: number analyzed (Participants) | 23 | 22
  Week 32; n=23, 22 | 90.0 (109.70) | 122.1 (122.65)
  Week 40; n=20, 15: number analyzed (Participants) | 20 | 15
  Week 40; n=20, 15 | 139.5 (82.72) | 137.1 (122.36)
  Week 48; n=7, 9: number analyzed (Participants) | 7 | 9
  Week 48; n=7, 9 | 125.0 (88.72) | 175.1 (64.64)
  Week 60; n=4, 2: number analyzed (Participants) | 4 | 2
  Week 60; n=4, 2 | 127.0 (99.39) | 158.5 (79.90)
  Week 72; n=1, 1: number analyzed (Participants) | 1 | 1
  Week 72; n=1, 1 | 0.0 (NA) — The standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 171.0 (NA) — The standard deviation could not be calculated as a single participant was analyzed at the specified time point.

10. Secondary Outcome: Change From Baseline in CD4+ Cell Count Over Time-Stage 2
Description: This end point was not evaluated in Stage 2 due to early termination of the study during Stage 1.
Time Frame: Baseline and up to Week 96
Population: mITT Population (observed). Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Percentage of CD4+ Cells Over Time-Stage 1
Description: The percentage of CD4+ cells was assessed using flow cytometry. Baseline is the last value on or before the start of study treatment. Change from Baseline was calculated as the value at specified visit minus the Baseline value. NA indicates data was not available. The standard deviation could not be calculated as a single participant was analyzed at the specified time point.
Time Frame: Baseline and up to Week 72
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of CD4+ cells
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 38 | 35
Percentage of CD4+ cells
  Week 4; n=37, 33: number analyzed (Participants) | 37 | 33
  Week 4; n=37, 33 | 1.94 (2.701) | 1.82 (2.152)
  Week 8; n=36, 30: number analyzed (Participants) | 36 | 30
  Week 8; n=36, 30 | 1.80 (2.495) | 1.69 (2.490)
  Week 12; n=35, 32: number analyzed (Participants) | 35 | 32
  Week 12; n=35, 32 | 3.41 (3.760) | 2.88 (3.084)
  Week 16; n=34, 31: number analyzed (Participants) | 34 | 31
  Week 16; n=34, 31 | 3.14 (3.486) | 3.66 (3.155)
  Week 24; n=31, 28: number analyzed (Participants) | 31 | 28
  Week 24; n=31, 28 | 4.71 (2.914) | 4.72 (3.315)
  Week 32; n=23, 22: number analyzed (Participants) | 23 | 22
  Week 32; n=23, 22 | 4.13 (3.671) | 4.81 (4.237)
  Week 40; n=20, 15: number analyzed (Participants) | 20 | 15
  Week 40; n=20, 15 | 5.38 (3.460) | 5.38 (3.318)
  Week 48; n=7, 9: number analyzed (Participants) | 7 | 9
  Week 48; n=7, 9 | 7.09 (4.271) | 7.16 (3.777)
  Week 60; n=4, 2: number analyzed (Participants) | 4 | 2
  Week 60; n=4, 2 | 7.95 (2.121) | 10.05 (2.616)
  Week 72; n=1, 1: number analyzed (Participants) | 1 | 1
  Week 72; n=1, 1 | 12.50 (NA) — The standard deviation could not be calculated as a single participant was analyzed at the specified time point. | 10.70 (NA) — The standard deviation could not be calculated as a single participant was analyzed at the specified time point.

12. Secondary Outcome: Change From Baseline in Percentage of CD4+ Cells Over Time-Stage 2
Description: This end point was not evaluated in Stage 2 due to early termination of the study during Stage 1.
Time Frame: Baseline and up to Week 96
Population: mITT Population (observed). Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events (AEs) Leading to Discontinuation (AELD)-Stage 1
Description: An SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or causes prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or medical events that may jeopardize the participant or require intervention (medical or surgical) to prevent one of the outcomes mentioned before. The number of participants with SAEs and AELDs are presented.
Time Frame: Up to Week 96
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 38 | 35
Participants
  SAEs | 4 | 3
  AELD | 2 | 1

14. Secondary Outcome: Number of Participants With SAEs and AELDs-Stage 2
Description: This end point was not evaluated in Stage 2 due to early termination of the study during Stage 1.
Time Frame: Up to Week 96
Population: mITT Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Occurrence of New Acquired Immunodeficiency Syndrome (AIDS) Defining Events-Stage 1
Description: The occurrence of new AIDS defining events that is, Centers for Disease Control (CDC) Class C events in participants is presented.
Time Frame: Up to Week 96
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 38 | 35
Participants | 1 | 0

16. Secondary Outcome: Number of Participants With Occurrence of New AIDS Defining Events-Stage 2
Description: This end point was not evaluated in Stage 2 due to early termination of the study during Stage 1.
Time Frame: Up to Week 96
Population: mITT Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Maximum Observed Concentration (Cmax) for BMS-955176-Stage 1
Description: The pharmacokinetic (PK) assessments were planned to be performed on PK Population, which comprised of all treated participants who had any available concentration-time data; however, it was not performed due to the early termination of the study in Stage 1.
Time Frame: Week 2 (pre-dose, 1, 2, 2.5, 3, 4, 4.5, 5, 6, 8, 12 hours post-dose and 24 hours [morning pre-dose])
Population: PK Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Cmax for BMS-955176-Stage 2
Description: This end point was not evaluated, as the resulting information would only have been needed to help confirm the dose for Stage 2 (which never opened due to the early termination of the study in Stage 1).
Time Frame: Week 2 (pre-dose, 1, 2, 2.5, 3, 4, 4.5, 5, 6, 8, 12 hours post-dose and 24 hours [morning pre-dose])
Population: PK Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) for BMS-955176-Stage 1
Description: PK assessments were planned to be performed; however, it was not performed due to the early termination of the study in Stage 1.
Time Frame: Week 2 (pre-dose, 1, 2, 2.5, 3, 4, 4.5, 5, 6, 8, 12 hours post-dose and 24 hours [morning pre-dose])
Population: PK Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Tmax for BMS-955176-Stage 2
Description: as for outcome 18
Time Frame: Week 2 (pre-dose, 1, 2, 2.5, 3, 4, 4.5, 5, 6, 8, 12 hours post-dose and 24 hours [morning pre-dose])
Population: PK Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Observed Plasma Concentration at the End of a Dosing Interval (Ctau) for BMS-955176-Stage 1
Description: as for outcome 19
Time Frame: Week 2 (pre-dose, 1, 2, 2.5, 3, 4, 4.5, 5, 6, 8, 12 hours post-dose and 24 hours [morning pre-dose])
Population: PK Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Ctau for BMS-955176-Stage 2
Description: as for outcome 18
Time Frame: Week 2 (pre-dose, 1, 2, 2.5, 3, 4, 4.5, 5, 6, 8, 12 hours post-dose and 24 hours [morning pre-dose])
Population: PK Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Observed Pre-dose Plasma Concentration (C0) for BMS-955176-Stage 1
Description: as for outcome 19
Time Frame: Week 2 (pre-dose, 1, 2, 2.5, 3, 4, 4.5, 5, 6, 8, 12 hours post-dose and 24 hours [morning pre-dose])
Population: PK Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: C0 for BMS-955176-Stage 2
Description: as for outcome 18
Time Frame: Week 2 (pre-dose, 1, 2, 2.5, 3, 4, 4.5, 5, 6, 8, 12 hours post-dose and 24 hours [morning pre-dose])
Population: PK Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Area Under the Concentration-time Curve in One Dosing Interval (AUC[Tau]) for BMS-955176-Stage 1
Description: as for outcome 19
Time Frame: Week 2 (pre-dose, 1, 2, 2.5, 3, 4, 4.5, 5, 6, 8, 12 hours post-dose and 24 hours [morning pre-dose])
Population: PK Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: AUC(Tau) for BMS-955176-Stage 2
Description: as for outcome 18
Time Frame: Week 2 (pre-dose, 1, 2, 2.5, 3, 4, 4.5, 5, 6, 8, 12 hours post-dose and 24 hours [morning pre-dose])
Population: PK Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Emergence of HIV Drug Resistance-Stage 1
Description: Emergence of drug resistance was planned to be assessed using the most current version of International AIDS Society-United States of America (IAS-USA); however, it was not assessed due to the early termination of the study in Stage 1.
Time Frame: Up to Week 96
Population: mITT Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 1: BMS-955176 120 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD | Stage 1: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Number of Participants With Emergence of HIV Drug Resistance-Stage 2
Description: This end point was not evaluated, as the resulting information would only have been needed to help assess the risk for Stage 2 (which never opened due to the early termination of the study in Stage 1).
Time Frame: Up to Week 96
Population: mITT Population. Data was not collected as no participants were enrolled in Stage 2 of the study.
Arm/Group | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from the start of study treatment until Week 96.
Description: AEs and SAEs were collected in Stage 1 in the modified intent to treat (mITT) Population. Data were not collected in Stage 2 as no participants were enrolled in Stage 2.
Groups:
- Stage 1: BMS955176+ATV/r+DTG: Participants were administered a once daily (QD) oral dose of 120 milligram (mg) BMS-955176 in combination with atazanavir boosted with ritonavir (ATV/r) 300/100 mg QD and dolutegravir (DTG) 50 mg QD for a duration of 96 weeks. The doses were administered in the morning with a meal.
- Stage 1: TDF+ATV/r+DTG: Participants were administered a QD oral dose of 300 mg tenofovir (TDF) in combination with ATV/r 300/100 mg QD and DTG 50 mg QD for a duration of 96 weeks. The doses were administered in the morning with a meal.
Arm/Group | Stage 1: BMS955176+ATV/r+DTG | Stage 1: TDF+ATV/r+DTG | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/35 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/38 | 3/35 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 32/38 | 24/35 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: BMS955176+ATV/r+DTG (N=38) | Stage 1: TDF+ATV/r+DTG (N=35) | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD (N=0) | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD (N=0) | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD (N=0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: BMS955176+ATV/r+DTG (N=38) | Stage 1: TDF+ATV/r+DTG (N=35) | Stage 2: BMS-955176 120 mg QD+ATV 400 mg QD+DTG 50 mg QD (N=0) | Stage 2: BMS-955176 180 mg QD+ATV 400 mg QD+DTG 50 mg QD (N=0) | Stage 2: TDF 300 mg QD+ATV/r 300/100 mg QD+DTG 50 mg QD (N=0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital dysplasia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 20 (31) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (3) | 5 (8) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Ocular icterus (Hepatobiliary disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin unconjugated increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-01-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT02386098/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT02386098/SAP_001.pdf